CLINICAL TRIAL: NCT05986019
Title: Evaluating the Effects of Transcranial Focused Ultrasound (tFUS) on Fronto-striatal Resting State Functional Connectivity in Healthy Individuals
Brief Title: Transcranial Focused Ultrasound (tFUS) Modulation of Reward Network
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00127562
Record Dates: First submitted 2023-07-31; First posted 2023-08-14 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Active or Sham tFUS
Who Masked: Participant
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tFUS (Experimental): tFUS will be administered within the MRI scanner. Participants receive two, 10-min sessions of active tFUS spread 10 min apart targeting the nucleus accumbens.
  Interventions: Device: transcranial focused ultrasound (tFUS)
- Sham tFUS (Sham Comparator): No ultrasound will be delivered to the participant during the experiment. Participants will not know or be told whether they are receiving active- or sham- tFUS.
  Interventions: Device: transcranial focused ultrasound (tFUS)

INTERVENTIONS:
Device: transcranial focused ultrasound (tFUS) — Transcranial focused ultrasound (tFUS) is a promising new technology that is both noninvasive and may be focally applied to deep brain targets. tFUS utilizes transducers which contain piezoelectric elements to produce pulses of ultrasonic waves that summate deep in the brain. Transcranial focused ultrasound (tFUS) uses a single transducer fixed in a head-worn apparatus on the scalp to produce ultrasonic waves deep into the brain.

SUMMARY:
Aim: Evaluate whether sonicating the Nucleus Accumbens (NAc) with transcranial focused ultrasound modifies functional connectivity between the NAc and the prefrontal cortex (PFC).

In this single visit, open-label pilot trial, we plan to evaluate whether transcranial focused ultrasound (tFUS), delivered to the nucleus accumbens (NAc) within the magnetic resonance imaging (MRI) scanner will impact resting state functional connectivity between the NAc and functionally connected brain regions like the prefrontal cortex (PFC) and the anterior cingulate cortex (ACC) in up to 10 healthy individuals.

HYPOTHESIS : tFUS will reduce prefrontal cortex (PFC)-NAc functional connectivity, in healthy individuals. We will investigate this hypothesis by administering tFUS within to MRI scanner to healthy individuals and conduct resting state functional neuroimaging before- and after the tFUS stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Have the capacity and ability to provide one's own consent and sign the informed consent document

Exclusion Criteria:

* Contraindicated for MRI.
* Any current or recent untreated medical, neurological, or psychiatric conditions
* Metal implant devices in the head, heart, or neck.
* History of brain surgery.
* History of myocardial infarction or arrhythmia, bradycardia.
* Personal or family history of seizure or epilepsy or personal use of medications that substantially reduce seizure threshold (e.g., olanzapine, chlorpromazine, lithium).
* Personal history of head injury, concussion, or self-report of moderate to severe traumatic brain injury.
* Individuals suffering from frequent/severe headaches.
* Individuals with a reported history of psychosis or mania, or individuals who are actively manic or psychotic.
* Regular or recent pain medication use
* Moderate to severe alcohol use (>3 drinks/day) or illicit substance use (urine confirmed).
* Persons who are pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2024-06-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina Institute of Psychiatry, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham tFUS: The sham sessions will include a transducer that is connected in a similar fashion to that of active tFUS, however the cable will not be plugged into the system, thus no ultrasound will be delivered to the participant. Participants will not know or be told whether they are receiving active- or sham- tFUS.
  transcranial focused ultrasound (tFUS): Transcranial focused ultrasound (tFUS) is a promising new technology that is both noninvasive and may be focally applied to deep brain targets. tFUS utilizes transducers which contain piezoelectric elements to produce pulses of ultrasonic waves that summate deep in the brain. Transcranial focused ultrasound (tFUS) uses a single transducer fixed in a head-worn apparatus on the scalp to produce ultrasonic waves deep into the brain.
Period: Overall Study
Arm/Group | Active tFUS | Sham tFUS
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tFUS | Sham tFUS | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10
Healthy Individuals [Count of Participants; unit: Participants] | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Resting State Functional Connectivity
Description: The main outcomes of this study are brain imaging related. Using a neuroimaging technique called resting state functional connectivity, which is a statistical dependence between time series of electro-physiological activity and (de)oxygenated blood levels in distinct regions of the brain. Modularity is measured on a -1 to 1 scale, with higher scores indicating stronger community structure, or a stronger tendency of clusters of brain regions to separate into distinct, highly interconnected networks with sparse connections across networks. The optimal modularity value depends on the context. For example, during complex tasks lower modularity is better, while during basic, automatic tasks higher modularity is better.
Time Frame: 24 minutes
Measure: Mean (Standard Error); unit: z value
Arm/Group | Active tFUS | Sham tFUS
Number analyzed (Participants) | 5 | 5
z value | 0.069 (0.088) | 0.160 (0.094)

ADVERSE EVENTS:
Time Frame: 2 months
Description: This study enrolled 10 participants by the end of the study, among which 5 participants received active tFUS and the other 5 participants received sham tFUS. 0 out of 5 participants in the active group and 0 out of 5 participants in the sham group were reported to have any adverse event.
Arm/Group | Active tFUS | Sham tFUS
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT05986019/Prot_001.pdf
  • Informed Consent Form (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/19/NCT05986019/ICF_000.pdf